CLINICAL TRIAL: NCT06657430
Title: A Study on the Preference of Risperidone Dosage Forms
Status: Recruiting | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-85
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Schizophrenia; Bipolar Affective Disorder; Autism Spectrum Disorder; Conduct Disorder; Mental Retardation
Keywords: risperidone; patch; cross-sectional study; preference
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Autism Spectrum Disorder; Conduct Disorder; Intellectual Disability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients and their caregivers: Patients (and their caregivers) with psychiatric disorders for which risperidone is indicated, including schizophrenia, bipolar disorder, autism spectrum disorder, conduct disorder, and mental retardation.

SUMMARY:
This study aimed to understand patients' needs and preferences for antipsychotic dosage forms.

DETAILED DESCRIPTION:
This study aims to understand patients' needs and preferences for antipsychotic dosage forms and to clarify the clinical value of patch-form antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia, bipolar disorder, autism spectrum disorder, mental retardation or their primary caregivers who voluntarily participate in the study.

Exclusion Criteria:

* Have difficulty reading and understanding Chinese or refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with schizophrenia, bipolar disorder, autism spectrum disorder, mental retardation or their primary caregivers who voluntarily participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients (and their caregivers) who prefer risperidone patch-form medicine | "through study completion, an average of 6 months
  The proportion of patients (and their caregivers) who preferred risperidone patch among the respondents in this study

SECONDARY OUTCOMES:
Factors related to patients' preference for risperidone patch-form medicines | through study completion, an average of 6 months
  Patients' evaluation of the importance of each advantage of risperidone patch in a self-made questionnaire (5-point Likert scale score)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No